CLINICAL TRIAL: NCT06778460
Title: Effect of Perioperative Continuous Intravenous Infusion of Esketamine and Lidocaine on Postoperative Chronic Pain and Long-term Survival in Patients Undergoing Hepatectomy
Brief Title: Effect of Esketamine and Lidocaine on Postoperative Chronic Pain and Long-term Survival in Patients Undergoing Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-451-2
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Chronic Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the anesthesiologist, data collectors, the physicians performing the follow-up, and data analysts will be blinded to the group allocation. Blinding will maintain until the completion of the final analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine-lidocaine group (Experimental): Patients received esketamine (0.25 mg/kg) and lidocaine (1.5 mg/kg) at the induction of anesthesia, followed by the continuous infusion of esketamine (0.02 mg/kg∙h) and lidocaine (1.5 mg/kg∙h) until the end of surgery. Postoperatively, the patients received two pumps. One pump delivered a fixed-rate infusion of lidocaine at 1.0 mg.kg-1.h-1 and esketamine at 0.02 mg.kg-1.h-1 infusion for 72 hours. Another PCIA device contained sufentanil 2 ug/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Interventions: Drug: Esketamine-lidocaine group
- Placebo group (Placebo Comparator): Patients received the same volume of normal saline instead of lidocaine and esketamine until the end of surgery. Postoperatively, the patients received two pumps. One pump was the same volume of normal saline instead of lidocaine and esketamine. Another PCIA device contained sufentanil 2 ug/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Interventions: Other: Placebo group

INTERVENTIONS:
Drug: Esketamine-lidocaine group — In the esketamine-lidocaine group, patients received esketamine (0.25 mg/kg) and lidocaine (1.5 mg/kg) at the induction of anesthesia, followed by the continuous infusion of esketamine (0.02 mg/kg∙h) and lidocaine (1.5 mg/kg∙h) until the end of surgery. Postoperatively, the patients received two pumps. One pump delivered a fixed-rate infusion of lidocaine at 1.0 mg.kg-1.h-1 and esketamine at 0.02 mg.kg-1.h-1 infusion for 72 hours. Another PCIA device contained sufentanil 2 ug/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Other Names: Trial group
  Arms: Esketamine-lidocaine group
Other: Placebo group — In the conventional analgesia group, patients received the same volume of normal saline instead of lidocaine and esketamine until the end of surgery. Postoperatively, the paitents received two pumps. One pump was the same volume of normal saline instead of lidocaine and esketamine. Another PCIA device contained sufentanil 2 ug/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Arms: Placebo group

SUMMARY:
This study is a further observation and follow-up of the patients enrolled in the registration number ChiCTR230007164430 to further evaluate the effect of long-term infusion of esketamine and lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing hepatectomy.

DETAILED DESCRIPTION:
This study is a further observation and follow-up of the patients enrolled in the registration number ChiCTR230007164430 to further evaluate the effect of long term infusion of esketamine and lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing hepatectomy. 304 patients with primary liver cancer who meet the inclusion criteria were included. According to the random number, the patients were divided into esketamine-lidocaine group and conventional analgesia group. In the esketamine-lidocaine group, patients received esketamine (0.25 mg/kg) and lidocaine (1.5 mg/kg) at the induction of anesthesia, followed by the continuous infusion of esketamine (0.02 mg/kg∙h) and lidocaine (1.5 mg/kg∙h) until the end of surgery. Postoperatively, the patients used 2 pumps. One pump delivered a fixed-rate infusion of lidocaine at 1.0 mg.kg-1.h-1 and esketamine at 0.02 mg.kg-1.h-1 infusion for 72 hours. Another PCIA device contained sufentanil 2 ug/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline. In the placebo group, the same volume of normal saline instead of lidocaine and esketamine will be administered. Numeric rating scale (NRS) is used to evaluate pain at rest and light activities at postoperative 24, 48, 72 hours. Follow-up after discharge includes chronic pain, the impact of chronic pain on quality of life, the relapse-free survival and overall survival from postoperative 3 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Scheduled for elective hepatectomy;
3. ASA grade I-III.

Exclusion Criteria:

1. Patients who have been intubated in the ICU following surgery and do not have a planned extubation within 6 hours postoperatively.
2. Patients with a body weight less than 40 kg or greater than 100 kg.
3. Patients with cardiac conduction system abnormalities (second- or third-degree atrioventricular block) or cardiac insufficiency (left ventricular ejection fraction < 50%).
4. Patients with severe hepatic insufficiency (alanine aminotransferase [ALT], aspartate aminotransferase [AST], or bilirubin levels more than 2.5 times the upper limit of normal) or renal insufficiency (creatinine clearance rate < 60 mL/min).
5. Patients with a known hypersensitivity to the investigational drug.
6. Patients with a history of long-term opioid abuse.
7. Patients who are unable to communicate effectively.
8. Patients with serious comorbid medical conditions, such as uncontrolled hypertension, coronary heart disease, intracranial vascular malformations, or acute asthma exacerbations.
9. Patients with a history of epilepsy or a history of manic episodes.
10. Pregnant or breastfeeding women.
11. Patients with glaucoma.
12. Patients with preoperative cognitive dysfunction, bipolar disorder, or other psychiatric disorders, including mental retardation.
13. Patients with primary liver cancer in conjunction with malignant tumors of other organs (such as lung, kidney, intestine, etc.), or those with clinical symptoms or imaging findings suggestive of distant metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic pain at 3 months postoperatively | 3 months postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience. The impact of chronic pain on the quality of life is also assessed by Brief Pain Inventory score.

SECONDARY OUTCOMES:
The incidence of chronic pain at 6 months and 1 year postoperatively | Up to 1 year postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience. The impact of chronic pain on the quality of life is also assessed by Brief Pain Inventory score.
Overall survival after surgery | Up to 5 years postoperatively
  Overall survival is defined as the time between the date from surgery to the date of death.
Recurrence-free survival after surgery | Up to 5 years postoperatively
  Postoperative re-examination is based on the diagnosis of enhanced CT, MRI, ultrasound or blood examination to determine whether the patient has recurrence and metastasis. Recurrence-free time refers to the time from surgery to tumor recurrence based on the above CT, MRI, etc.
Disability-free surviva survival | Up to 5 years postoperatively
  Patient self-assessment is carried out by using the World Health Organization(WHO) Disability Scale, with a minimum score of 12 points and a maximum score of 60 points. The lower the score, the higher the quality of life.
The prevalence of neuropathic pain | Up to 1 year postoperatively
  The ID Pain scale is used as a validated assessment of neuropathic pain. ID pain questionnaire consists of six items.
  Pain higher scores suggest a neuropathic component to the pain.
Brief Pain Inventory(BPI) pain interference subscale score | Up to 1 year postoperatively
  BPI pain interference subscale is a 7-item questionnaire asking participants to describe how pain has interfered general activity, mood, walking, normal work, relations with others, sleep, and enjoyment of life. Each question is answered on a scale 0(does not interfere) to 10(completely interferes). The total range of score is 0-70. The higher the scores suggest the worse the interference.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China